CLINICAL TRIAL: NCT04547257
Title: Safety and Effectiveness Evaluation of Seraph 100 Microbind Affinity Blood Filter (Seraph 100) in the Treatment of Patients With COVID-19
Brief Title: Safety & Effectiveness Evaluation of Seraph 100 in Treatment of Pts With COVID-19
Acronym: CP022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ExThera Medical Europe BV (Industry)
Collaborators: ExThera Medical Corporation (Industry); Vivantes Clinic Neukölln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP022
Record Dates: First submitted 2020-04-29; First posted 2020-09-14 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The primary objective is to demonstrate the safety and effectiveness of the Exthera Medical Seraph 100 Microbind Affinity Blood Filter in the clinical improvement of SARS-CoV-2 infected patients, measured by the reduction of established and suspected prognostic parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Extracorporeal therapy with Seraph 100 blood filter
  Interventions: Device: Seraph 100
- Control (No Intervention): patients receive antibiotics only as standard of care

INTERVENTIONS:
Device: Seraph 100 — Bloodfiltration with Seraph 100
  Arms: Treatment

SUMMARY:
Safety and Effectiveness Evaluation of Seraph 100 Microbind Affinity Blood Filter (Seraph 100) in the treatment of patients with COVID-19

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, controlled clinical investigation designed to evaluate the safety and effectiveness of the Exthera Medical Seraph 100 Microbind Affinity Blood Filter in the treatment of patients with confirmed SARS-CoV-2 infection.

The clinical investigation will be conducted at 3 centers in Germany and at 2 centers in Spain. Subjects will be randomized to the treatment group (Seraph 100 + standard of care) versus control group (standard of care only).

Subjects will be followed for 28 days. For viral quantification, study-related serum samples are done immediately before the initial treatment with Seraph 100 starts in the treatment group or immediately after randomization into the control group. Additionally, serum sampling at timepoint 12 hours is applicable for both treatment and control group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with confirmed SARS-CoV-2 infection
2. Be ≥ 18 years old and ≤90 years old
3. Acute respiratory distress syndrome assessed by a modified Sequential Organ Failure Assessment score of at least 2 points
4. At least one additional organ dysfunction assessed by a modified Sequential Organ Failure Assessment score of at least 1 point
5. Written or electronic consent of the subjects who are legally competent and have the capacity to give consent

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
3. Presence of comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
4. Have Child-Pugh Class C cirrhosis
5. Have platelet count <30.000/uL
6. Contraindications for heparin sodium for injection
7. Subjects demonstrating any contraindication for this treatment as described in the IFU
8. Subjects with known allergy of polyethylene and copolyester
9. Subjects with hospital-acquired SARS-CoV-2 infections
10. Subject is held in an institution by court or official order
11. Subject is dependent on the sponsor or investigator so that consent can no longer be considered voluntary

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Organ failure | 48 hours after initial treatment
  Change in organ failure as assessed by a modified Sequential Organ Failure Assessment score (range, 0-20, with higher scores indicating more dysfunction) from baseline to 48 hours

SECONDARY OUTCOMES:
Change in Organ Failure | Daily during ICU stay from the start of the initial treatment until day 4
  Change in organ failure as assessed by a modified Sequential Organ Failure Assessment score (range 0 - 20, with higher scores indicating more dysfunction)
All-cause mortality | 28 days
  All-cause mortality
Organ dysfunction-free days | Daily during ICU stay (up to 28 days)
  Organ dysfunction-free days
Intensive Care Unit (ICU) complications | Daily during ICU stay (up to 28 days)
  Intensive Care Unit (ICU) complications
Ventilator-free days (VFDs) | Daily during ICU stay (up to 28 days)
  Ventilator-free days (VFDs)
Length of stay (LOS) at ICU and hospital ward | During ICU and hospital ward stay (up to 28 days)
  Length of stay (LOS) at ICU and hospital ward
Prognosis Factors | From baseline up to 48 hours
  Prognosis factors (D-Dimer, Troponin T, Ferritin, NTpro-BNP, LDH, IL6, sIL2)
Recurrence of sepsis | 7 days
  Recurrence of sepsis
Persistence of sepsis | 7 days
  Persistence of sepsis

OTHER OUTCOMES:
N (%) of patients with treatment emergent adverse events | Occurrence within the 28 days follow-up period
  N (%) of patients with treatment emergent adverse events
Laboratory data | Daily during ICU stay (up to 28 days)
  Laboratory data (blood test, hematology, chemistry, coagulation, and blood gases)
Vital signs score | Daily during ICU stay (up to 28 days)
  Vital signs score
Physical examination score | Daily during ICU stay (up to 28 days)
  Physical examination score
Reduction of viral load | During treatment (minimum treatment duration is 5 hours, maximum treatment duration is 24 hours)
  Reduction of viral load

CONTACTS AND LOCATIONS:
Overall Officials: Herwig Gerlach, Prof., Principal Investigator — Vivantes Neukoelln Berlin
Locations (5):
- Germany (3):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Vivantes Klinikum Neukölln, Berlin
  - Universitätsklinikum Essen, Essen
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will be responsible for determining whether to register the clinical investigation on www.clinicaltrials.gov or any other clinical trials, in accordance with the International Committee of Medical Journal Editors guidelines, or any other applicable guidelines.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: in 9 months
URL: http://extheramedical.com